CLINICAL TRIAL: NCT04524091
Title: Inspiratory Ratio: Predictor of Inspiratory Effort Response to High Positive End Expiratory Pressure in Patients Recovering From Acute Respiratory Distress Syndrome.
Brief Title: Inspiratory Ratio: Predictor of Inspiratory Effort Response to High PEEP in Patients Recovering From ARDS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sanatorio Anchorena San Martin (Other)
Responsible Party: Principal Investigator, Matias Accoce, Head of physica therapy department, Sanatorio Anchorena San Martin
Other Study IDs: 20.2020
Record Dates: First submitted 2020-08-19; First posted 2020-08-24 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Positive-Pressure Respiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Positive end expiratory pressure — Initially, the patients will be ventilated using pressure support ventilation with an inspiratory pressure adjusted to achieve 6 - 8 ml/kg of PBW with a minimal esophageal pressure swing of 5 cmH2O and a PEEP of 5 cmH2O. After 5 minutes, we will measure five IPSexp and five IPSinsp in random order and considering a resting period between each occlusion in order to avoid learning effect and disconfort. The IR will be calculated using the average of the measured IPSexp and the average of the IPSinsp. Besides, we will register the average of esophageal pressure and transpulmonary pressure swings continuously. The same procedure will be carried out with 10 and 15 cmH2O of PEEP. Inspiratory pressure will be kept constant throughout the protocol.

SUMMARY:
Spontaneous Breathing (SB) can be potentially harmful in patient with Acute Respiratory Distress Syndrome (ARDS) during the transition phase of passive ventilation to partial ventilatory support. The application of high Positive End Expiratory Pressure (PEEP) during SB has shown to ameliorate the progression of lung injury by decreasing the TP and esophageal pressure (EP) swings and the stress / strain applied to the lung. The mechanisms proposed to be responsible for these effects are the activation of Hering Breuer reflex, the recruitment of previously collapsed tissue, the homogenization of lung and the improvement of respiratory system compliance and the impairment in the length - tension relationship of the diaphragm. If all the previously explained mechanisms have an effect on the control of inspiratory effort, a decrease in the intensity of effort is expected during an end-inspiratory occlusion in patients who will respond to high PEEP application. Based on this rationale, the investigators developed an index called "Inspiratory Ratio" (IR) to predict the response of patient's inspiratory effort to the application of high PEEP without need of esophageal manometry.

DETAILED DESCRIPTION:
Spontaneous Breathing (SB) can be potentially harmful in patient with Acute Respiratory Distress Syndrome (ARDS) during the transition phase of passive ventilation to partial ventilatory support. A high respiratory drive and consequently, a strong inspiratory effort, may produce large transpulmonary pressure (TP) swings mainly in dependent lung regions closer to the diaphragm and cause alveolar rupture and inflammatory mediators release.

The application of high Positive End Expiratory Pressure (PEEP) during SB has shown to ameliorate the progression of lung injury by decreasing the TP and esophageal pressure (EP) swings and the stress / strain applied to the lung. The mechanisms proposed to be responsible for these effects are the activation of Hering Breuer reflex caused by a greater stretch of the lung parenchyma at the end of inspiration; the recruitment of previously collapsed tissue, the homogenization of lung ("fluid like behavior") and the improvement of respiratory system compliance (Crs); and the impairment in the length - tension relationship of the diaphragm which produces mechanical disadvantage to generate force due to a higher lung volume. However, it is uncertain which patient will respond adequately to the application of high PEEP and consequently will reduce the inspiratory effort.

If all the previously explained mechanisms have an effect on the control of inspiratory effort, in patients who will respond to high PEEP application, a decrease in inspiratory effort is expected during an end-inspiratory occlusion. At end-inspiration lung parenchyma is more homogeneous, the lung volume is higher and the diaphragmic dome is flatter compared to the physiological condition end of expiration, where the lung volume is lower, the parenchyma is more heterogeneous and the diaphragmatic neuromechanical coupling is better. Based on this rationale, the investigators developed an index called "Inspiratory Ratio" (IR) to predict the response of patient's inspiratory effort to the application of high PEEP without having to measure esophageal pressure.

The IR will be calculated using the following formula: (IPSexp - IPSinsp ) / (IPSexp) x 100

IPSexp = negative deflection in airway pressure expiratory pause; IPSinsp = negative deflection in airway pressure end inspiratory pause

ELIGIBILITY:
Inclusion Criteria:

* Need of invasive mechanical ventilation
* Patients who had fulfill ARDS criteria based on Berlin definition during any time of invasive mechanical ventilation.
* Patient ventilated in pressure support ventilation.
* Time of invasive ventilation expected to be longer than 24 hs after the day of enrollment.

Exclusion Criteria:

* Neuromuscular diseases (e.g., amyotrophic lateral sclerosis, Duchenne Erb)
* previous diagnosis of chronic obstructed pulmonary disease
* not resolved pneumothorax
* bronchopleural fistula
* suspicion of central respiratory drive alteration (e.g., benzodiazepines intoxication).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute respiratory distress syndrome ventilated using an endotracheal tube admitted to Anchorena San Martin intensive care unit who are ventilated in pressure support ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Inspiratory ratio | 10 minutes
  Inspiratory ratio will be calculated using the formula (IPSexp - IPSinsp )/IPSexp x 100, being IPSexp = negative deflection in airway pressure during an end expiratory pause; IPSinsp = negative deflection in airway pressure during an end inspiratory pause.

SECONDARY OUTCOMES:
Esophageal pressure swing | 10 minutes
  Esophageal pressure swing will be calculated as the difference between end expiration and end inspiration esophageal pressure during the las 30-60 seconds of each PEEP condition evaluated
Dynamic transpulmonary pressure swing | 10 minutes
  Dynamic transpulmonary pressure swing will be calculated as the difference between end expiration and end inspiration dynamic transpulmonary pressure during the las 30-60 seconds of each PEEP condition evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Sanatorio Anchorena de San Martin, San Martín, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Esteban A, Frutos-Vivar F, Muriel A, Ferguson ND, Penuelas O, Abraira V, Raymondos K, Rios F, Nin N, Apezteguia C, Violi DA, Thille AW, Brochard L, Gonzalez M, Villagomez AJ, Hurtado J, Davies AR, Du B, Maggiore SM, Pelosi P, Soto L, Tomicic V, D'Empaire G, Matamis D, Abroug F, Moreno RP, Soares MA, Arabi Y, Sandi F, Jibaja M, Amin P, Koh Y, Kuiper MA, Bulow HH, Zeggwagh AA, Anzueto A. Evolution of mortality over time in patients receiving mechanical ventilation. Am J Respir Crit Care Med. 2013 Jul 15;188(2):220-30. doi: 10.1164/rccm.201212-2169OC. PMID 23631814
- [Background] DAS-Taskforce 2015; Baron R, Binder A, Biniek R, Braune S, Buerkle H, Dall P, Demirakca S, Eckardt R, Eggers V, Eichler I, Fietze I, Freys S, Frund A, Garten L, Gohrbandt B, Harth I, Hartl W, Heppner HJ, Horter J, Huth R, Janssens U, Jungk C, Kaeuper KM, Kessler P, Kleinschmidt S, Kochanek M, Kumpf M, Meiser A, Mueller A, Orth M, Putensen C, Roth B, Schaefer M, Schaefers R, Schellongowski P, Schindler M, Schmitt R, Scholz J, Schroeder S, Schwarzmann G, Spies C, Stingele R, Tonner P, Trieschmann U, Tryba M, Wappler F, Waydhas C, Weiss B, Weisshaar G. Evidence and consensus based guideline for the management of delirium, analgesia, and sedation in intensive care medicine. Revision 2015 (DAS-Guideline 2015) - short version. Ger Med Sci. 2015 Nov 12;13:Doc19. doi: 10.3205/000223. eCollection 2015. PMID 26609286
- [Background] Schepens T, Dres M, Heunks L, Goligher EC. Diaphragm-protective mechanical ventilation. Curr Opin Crit Care. 2019 Feb;25(1):77-85. doi: 10.1097/MCC.0000000000000578. PMID 30531536
- [Background] Mauri T, Cambiaghi B, Spinelli E, Langer T, Grasselli G. Spontaneous breathing: a double-edged sword to handle with care. Ann Transl Med. 2017 Jul;5(14):292. doi: 10.21037/atm.2017.06.55. PMID 28828367
- [Background] Goligher EC, Fan E, Herridge MS, Murray A, Vorona S, Brace D, Rittayamai N, Lanys A, Tomlinson G, Singh JM, Bolz SS, Rubenfeld GD, Kavanagh BP, Brochard LJ, Ferguson ND. Evolution of Diaphragm Thickness during Mechanical Ventilation. Impact of Inspiratory Effort. Am J Respir Crit Care Med. 2015 Nov 1;192(9):1080-8. doi: 10.1164/rccm.201503-0620OC. PMID 26167730
- [Background] Telias I, Brochard L, Goligher EC. Is my patient's respiratory drive (too) high? Intensive Care Med. 2018 Nov;44(11):1936-1939. doi: 10.1007/s00134-018-5091-2. Epub 2018 Mar 1. No abstract available. PMID 29497778
- [Background] Brochard L, Slutsky A, Pesenti A. Mechanical Ventilation to Minimize Progression of Lung Injury in Acute Respiratory Failure. Am J Respir Crit Care Med. 2017 Feb 15;195(4):438-442. doi: 10.1164/rccm.201605-1081CP. PMID 27626833
- [Background] Morais CCA, Koyama Y, Yoshida T, Plens GM, Gomes S, Lima CAS, Ramos OPS, Pereira SM, Kawaguchi N, Yamamoto H, Uchiyama A, Borges JB, Vidal Melo MF, Tucci MR, Amato MBP, Kavanagh BP, Costa ELV, Fujino Y. High Positive End-Expiratory Pressure Renders Spontaneous Effort Noninjurious. Am J Respir Crit Care Med. 2018 May 15;197(10):1285-1296. doi: 10.1164/rccm.201706-1244OC. PMID 29323536
- [Background] Yoshida T, Uchiyama A, Matsuura N, Mashimo T, Fujino Y. Spontaneous breathing during lung-protective ventilation in an experimental acute lung injury model: high transpulmonary pressure associated with strong spontaneous breathing effort may worsen lung injury. Crit Care Med. 2012 May;40(5):1578-85. doi: 10.1097/CCM.0b013e3182451c40. PMID 22430241
- [Background] Mauri T, Bellani G, Confalonieri A, Tagliabue P, Turella M, Coppadoro A, Citerio G, Patroniti N, Pesenti A. Topographic distribution of tidal ventilation in acute respiratory distress syndrome: effects of positive end-expiratory pressure and pressure support. Crit Care Med. 2013 Jul;41(7):1664-73. doi: 10.1097/CCM.0b013e318287f6e7. PMID 23507723